CLINICAL TRIAL: NCT03399071
Title: Study Title: Peri-operative Immuno-Chemotherapy in Operable Oesophageal and Gastric Cancer (ICONIC Trial)
Brief Title: Study Title: Peri-operative Immuno-Chemotherapy in Operable Oesophageal and Gastric Cancer
Acronym: ICONIC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4557
Record Dates: First submitted 2017-11-16; First posted 2018-01-16 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Gastric Adenocarcinoma; Oesophageal Adenocarcinoma
Keywords: Gastric cancer; Oesophageal cancer; Gastro-oesophageal cancer; Perioperative; Immunotherapy; Anti PDL1; Avelumab; FLOT
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Stomach Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients will receive chemo-immunotherapy consisting of FLOT chemotherapy and the PD-L1 inhibiting monoclonal antibody Avelumab. Four cycles of two-weekly chemo-immunotherapy will be administered before surgery and four further cycles post-operatively in patients who are fit enough to receive further chemo-immunotherapy after surgery. Resectional surgery will take place 4-8 weeks following the last dose of chemo-immunotherapy in patients who remain fit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FLOT plus Avelumab (FLOT-A) (Experimental): Avelumab 10mg/kg (or Maximum Administered Dose established in safety run-in) iv infusion over 1 hour.
  Followed by FLOT: Oxaliplatin 85mg/m2 iv infusion day 1 over 2 hours, Folinic acid 200mg/m2 iv infusion day 1 over 2 hours, Docetaxel 50mg/m2 iv day 1 over 1 hour, Fluorouracil 2600mg/m2 over 24 hours iv
  Interventions: Drug: FLOT-A

INTERVENTIONS:
Drug: FLOT-A — This is a single-arm study with all patients receiving combination FLOT-A

SUMMARY:
A single centre phase II trial of peri-operative chemo-immunotherapy in operable gastro-oesophageal adenocarcinoma (GOA). This trial is designed to evaluate the safety and efficacy of administering Avelumab, an anti-PD-L1 monoclonal antibody, with cytotoxic FLOT chemotherapy for patients with operable GOA treated according to a peri-operative protocol.

This trial is in 2 stages: the first stage will establish the safe and tolerated maximum administered dose (MAD) of Avelumab in combination with FLOT and the second stage will assess the efficacy of this combination therapy in achieving pathological complete response (pCR) and peri-operative safety.

DETAILED DESCRIPTION:
Patients will receive chemo-immunotherapy consisting of FLOT chemotherapy (Folinic acid 200mg/m2 iv infusion day 1, Oxaliplatin 85mg/m2 iv infusion day 1, Docetaxel 50mg/m2 iv day 1, Fluorouracil 2600mg/m2 over 24 hours iv) and the PD-L1 inhibiting monoclonal antibody Avelumab. The safe dose of Avelumab in combination with FLOT will be established in a safety run-in phase with a standard 3+3 design, starting with the recommended dose of 10mg/kg iv Avelumab (dose level 0) in which a dose reduction to 7mg/kg iv (dose level -1) may occur. Four cycles of two-weekly chemo-immunotherapy will be administered before surgery and four further cycles post-operatively in patients who are fit enough to receive further chemo-immunotherapy after surgery. Resectional surgery will take place 4-8 weeks following the last dose of chemo-immunotherapy in patients who remain fit.

Study Objectives:

To evaluate the safety, efficacy and toxicities and to explore biomarkers of peri-operative chemo-immunotherapy with Avelumab and FLOT.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female patients aged ≥18 years
2. Histologically confirmed gastric, gastro-oesophageal junction or oesophageal adenocarcinoma (referred to as gastro-oesophageal adenocarcinoma (GOA) in this protocol).
3. Oesophageal and gastric tumours should be TNM7 stage T1-4 and N0-N2, with no evidence of distant metastases (M0) where the MDT believes that an R0 resection can be achieved after pre-operative chemotherapy.
4. Absence of distant metastases on CT scan and PET scan and staging laparoscopy (where indicated) prior to study entry
5. No prior therapy for GOA
6. Considered fit for surgery by surgical/anaesthetic team
7. Adequate bone marrow function:

   * Absolute neutrophil count (ANC) >1.5x10-9/L
   * White blood count >3x10-9/L
   * Platelets ≥100x10-9/L
   * Haemoglobin (Hb) >9g/dL (can be post-transfusion)
8. Adequate renal function: Creatinine Clearance of >50ml/min or measured EDTA Clearance of ≥50ml/min. If the calculated Creatinine Clearance is <60ml/min then a measured EDTA Clearance is required. If available, the EDTA Clearance should always take precedence over the Creatinine Clearance.
9. Adequate liver function

   * Serum bilirubin <22 umol/L
   * ALT/AST ≤2.5x ULN
10. Adequate coagulation profile

    * International Normalised Ratio (INR) < 1.5
    * Activated Prothrombin Time (APTT) < 1.5xULN
11. Patients on oral anticoagulation are advised to change to low molecular weight heparin prior to study entry, to be eligible
12. ECOG performance status 0 or 1
13. Body Mass Index (BMI) ≤30
14. Patient is fit to undergo all protocol investigations and receive all protocol treatment based on the assessment in the surgical and oncology clinics. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrolment.
15. Willingness and ability to comply with the protocol for the duration of the study including scheduled visits, examinations, investigations and treatment plans

Exclusion Criteria

Patients are not eligible for the trial if any of the exclusion criteria below are met:

1. Any contraindication or known hypersensitivity reaction to any of the study drugs, or components of Folinic acid, Oxaliplatin, 5FU or Docetaxel
2. Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 NCI CTCAE v 4.0), any history of anaphylaxis, or uncontrolled asthma (i.e., 3 or more features of partially controlled asthma)
3. If known dihydropyrimidine dehydrogenase (DPD) deficiency, patients must be deemed safe to receive appropriate dose-adjusted 5-FU according to the identified mutation.
4. Patients who have received anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
5. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
6. Patients recommended to have radiotherapy as part of routine management for their GOA are ineligible
7. Any immunodeficiency disorder
8. Any active autoimmune disease that has required systemic treatment in the past 2 years (i.e, with use of disease modifying agents, corticosteroids or immunosuppressive drugs) or is expected to deteriorate when receiving avelumab, with the following exceptions:

   * Patients only receiving hormone replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy (doses ≤10mg - or equivalent - of prednisolone per day) for adrenal or pituitary insufficiency) are eligible.
   * Patients with vitiligo or psoriasis not requiring immunosuppressive treatment are eligible
   * Patients requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement
   * Administration of steroids through a route known to result in minimal systemic exposure (topical, intranasal intra-ocular, or inhalation) are acceptable. Steroids as pre-medication for hypersensitivity reactions e.g. CT contrast are also acceptable
9. Prior organ transplantation, including allogeneic stem-cell transplantation
10. History of inflammatory bowel disease with the following exception:

    • Patients with a history of ulcerative colitis who have had a colectomy are eligible
11. Patients with a history of interstitial lung disease or radiological evidence of pulmonary fibrosis
12. Cerebrovascular disease (including transient ischaemic attacks (TIA) and strokes) within the previous year
13. Cardiovascular diseases as follows:

    * Myocardial infarction within the previous year
    * Serious cardiac arrhythmia requiring medication (for example, ventricular tachycardia, supraventricular tachycardia or atrial fibrillation with a resting heart rate > 110bpm)
    * Unstable angina
    * Congestive cardiac arrhythmia (New York Heart Association Classification Class II or above)
14. Other severe acute or chronic medical conditions or psychiatric conditions including recent (within the past year) active suicidal ideation or behaviour
15. Current signs or symptoms of any other severe progressive or uncontrolled hepatic, haematologic, gastrointestinal, endocrine, respiratory or cardiac disease other than directly related to gastrooesophageal adenocarcinoma, which in the opinion of the investigator,might impair the subject's tolerance of trial treatment or procedures.
16. Major surgery, major trauma or open biopsy within 28 days prior to registration (not including staging laparoscopy)
17. Evidence of bleeding diathesis or coagulopathy
18. Active infection requiring systemic therapy, non-healing wound, ulcer or bone fracture requiring therapy
19. Known positive tests for human immunodeficiency virus (HIV) infection
20. Active Hepatitis A, B or C infection. If there is a previous history of Hepatitis infection which has been treated and cleared, there must be evidence that disease is not currently active.
21. Known peripheral neuropathy > grade 1 (absence of deep tendon reflexes as the sole neurological abnormality does not render the patient ineligible)
22. Use of live attenuated vaccine within 28 days of initiation of study therapy, or anticipation that a live attenuated vaccine will be required during the study
23. Pregnancy/of child bearing potential. Pregnancy must be excluded with a negative serum pregnancy test, within 7 days before initiation of therapy, if the risk of conception exists. Sexually active female patients must be surgically sterile or be postmenopausal or must agree to use highly effective contraception. Sexually active male patients must be surgically sterile or must agree to use highly effective contraception, i.e. methods with a failure rate of <1% per year (see section 5.4 for full definition and examples of highly effective contraception). Lactation- breast-feeding is contraindicated and must be discontinued for the duration of the trial and for at least 1 month afterward the last dose of Avelumab.
24. Any patient specific factors which are likely to interfere with compliance of trial specific procedures or treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate of combination FLOT-A | Within 2 years of study opening
  The primary objective is to assess the efficacy of FLOT-A in the peri-operative setting in patients with operable GOAs. We aim to increase the pCR rate after peri-operative treatment from 10% (minimum expected path CR rate for peri-operative FLOT chemotherapy), to a superior pCR rate of >25%, by adding Avelumab to FLOT.
  Complete histopathologic response is defined by no vital tumour cells neither in the oesophagus, the stomach nor in the regional lymph nodes. In cases of residual tumour, the response assessment will follow criteria described by Mandard et al.

SECONDARY OUTCOMES:
Number of participants with grade 3 or 4 treatment-related adverse events as assessed by CTCAE v4.0 | Within 2 years
  Safety of peri-operative FLOT-A will be assessed by summarising grade 3-4 toxicity and DLT rates as proportions.
Radiological response rate using RECIST 1.1 criteria | Within 3 years
  Radiological response rate assessed at the pre-operative scan using RECIST 1.1 criteria. Radiological tumour response before surgery will be defined as partial response or complete response.
Median progression free survival by Kaplan Meir method | Within 5 years
  PFS will be summarised using Kaplan Meier methods, presenting median survival with 95% confidence intervals. PFS is defined as time from registration to clinical/radiological progression or death from any cause. Patients event free at time of analysis will be censored at last follow-up date.
Median overall survival by Kaplan Meir method | Within 5 years
  OS will be summarised using Kaplan Meier method, presenting median survival with 95% confidence intervals. OS is defined as time from registration to date of death of any cause. Patients event free at time of analysis will be censored at last follow-up date.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Gerlinger, MD, FRCP, Principal Investigator — The Royal Marsden NHSFT
Locations (1):
- The Royal Marsden Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang X, Ge X, Zhang Y, Xue X. The current management and biomarkers of immunotherapy in advanced gastric cancer. Medicine (Baltimore). 2022 May 27;101(21):e29304. doi: 10.1097/MD.0000000000029304. PMID 35623069